CLINICAL TRIAL: NCT04187794
Title: Assessment of the Literacy Level of Patients With Chronic Rheumatic Diseases and Association With the Level of Knowledge and Medication Adherence: For a Better Integration of Patients' Literacy Levels Into Their Therapeutic Management.
Brief Title: Rheumatic Diseases: Evaluation of Health LIteracy, Medication adhereNce and Knowledges
Acronym: LINK
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0746
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Rheumatic Diseases; Treatment Adherence
MeSH Terms: conditions — Rheumatic Diseases; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Interview patient — to investigate an association between literacy level and medication adherence in patients with rheumatic diseases.

SUMMARY:
A medication non-adherence is reported in chronic rheumatic diseases, in a context of complex and long-term treatments (injectable/per os targeted therapies, biosimilar...). Understanding and integrating the patient into a shared medical decision are key factors for adherence. From this perspective, the level of literacy (an individual's ability to find, understand and use health information) must be explored in order to adapt the communication of information. These are currently insufficiently adapted to the individual understanding of patients. In practice, literacy assessment is very poorly integrated into routine care, while several tools are validated in French. In rheumatology, foreign studies have shown that literacy is positively related to knowledge level. The results remain contradictory regarding its association with medication adherence. Today, the literacy level of patients with rheumatic diseases and its impact on adherence has not been studied in France, although these evaluations would be useful to adapt interventions individually. The acceptance of patients to complete a literacy assessment questionnaire during their care should also be analysed as a condition of its deployment.

ELIGIBILITY:
Inclusion Criteria:

* patient older than 18 years
* Having at least 6 months of disease-modifying rheumatic treatment (methotrexate and/or targeted treatment (anti-JAK) and/or subcutaneous biotherapies)
* Understanding French,
* With good visual acuity.

Exclusion Criteria:

* Patients with cognitive disorders
* Pregnant, parturient and lactating women
* Persons deprived of their liberty
* Major persons who are subject to a legal protection measure (guardianship, curators)
* Persons not affiliated to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a rheumatic disease (rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis) hospitalized (conventional or day hospitalization) or in consultation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Correlation between Literacy and medication levels | At inclusion
  Correlation coefficient between literacy level (HLS-EU-16: European Health Literacy scale) and medication adherence level (CQR: Compliance Questionnaire Rheumatology).

CONTACTS AND LOCATIONS:
Overall Officials: Anne Laure YAILIAN, PD, Principal Investigator — Service hospitalier de rhumatologie
Locations (1):
- Service de rhumatologie Hôpital Edouard Herriot, Lyon, France